CLINICAL TRIAL: NCT01132417
Title: In Vitro Activity of Tigecycline Among Key Bacterial Pathogens Exhibiting Multidrug Resistance
Status: Suspended | Type: Observational
Why Stopped: researchers delay
Sponsor: King Faisal University (Other)
Responsible Party: Wyeth Pharmaceuticals FZ-LLC, Middle East and North America Region, King Faisal University
Other Study IDs: 3074X1-4548
Record Dates: First submitted 2009-09-19; First posted 2010-05-28 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Infections, Bacterial
Keywords: Tigecycline, MDR; Patient infected with multidrug resistance bacteria
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum, whole blood, urine, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multidrug resistant (MDR)bacterial strains
  Interventions: Drug: In Vitro activity of Tigecycline among key bacterial pathogens exhibiting multidrug resistance

INTERVENTIONS:
Drug: In Vitro activity of Tigecycline among key bacterial pathogens exhibiting multidrug resistance — studies in human beings in which biomedical and/or health outcomes are assessed in pre-defined groups of individuals. Subjects in the study may receive diagnostic, therapeutic, or other interventions, but the investigator does not assign specific interventions to the subjects of the study.

SUMMARY:
Observational: studies in human beings in which biomedical and/or health outcomes are assessed in pre-defined groups of individuals. Subjects in the study may receive diagnostic, therapeutic, or other interventions, but the investigator does not assign specific interventions to the subjects of the study.

DETAILED DESCRIPTION:
Study Phase Definition: Phase of investigation, as defined by the US FDA for trials involving investigational new drugs. Select only one.

N/A: for trials without phases Observational Study Design Case-control: group of individuals with specific characteristics (e.g., conditions or exposures) compared to group(s) with different Time Perspective Cross-sectional: observations or measurements made at a single point in time, usually at subject enrollment Biospecimen Retention - select one Samples Without DNA - samples retained, with no potential for DNA extraction from any retained samples (e.g., fixed tissue, plasma) Biospecimen Description

Sputum, whole blood, urine, tissue Enrollment

Single group study Number of Groups/Cohorts Definition: Number of study groups/cohorts. Enter 1 for a single-group study. Many observational studies have one group/cohort; case control studies typically have two.

One study group, anticipated samples in the rang of 400-500 samples 8. Arms, Groups and Interventions N/L Group/Cohort Label

ELIGIBILITY:
Inclusion Criteria:

* All patients with infection with MDRs infections will be included

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Definition: For observational studies only, a description of the population from which the groups or cohorts will be selected (e.g., primary care clinic, community sample, residents of a certain town).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Asim E Ltayeb Diab, MD, Ph D, Principal Investigator — Assist. Professor and Consultant Microbiologist
Locations (1):
- King Faisal Univrsity, Departmentof Microbiology and Immunology,, dammam branh, Dammam, Eastern Province, Saudi Arabia